CLINICAL TRIAL: NCT07356791
Title: Phase II Prospective Cohort Study of Intravesical Recombinant Human Type 5 Adenovirus Injection for Treatment of High-Risk Non-Muscle Invasive Bladder Cancer: Evaluating Efficacy and Safety (REBIRTH-013)
Brief Title: Phase II Prospective Cohort Study of Intravesical Recombinant Human Type 5 Adenovirus Injection for Treatment of High-Risk Non-Muscle Invasive Bladder Cancer: Evaluating Efficacy and Safety
Acronym: REBIRTH-013
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2024-0218
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer
Keywords: High-risk non-muscle invasive bladder cancer (HR-NMIBC); Bladder carcinoma in situ (CIS); Intravesical adenovirus therapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: The administration cycle of this experiment includes 6 induction perfusion periods (once a week for 6 consecutive weeks) and 15 maintenance perfusion periods (once a week for the first 3 weeks after 3, 6, 12, 18, and 24 months of initial induction perfusion, for a total of 3 times a month). This study will adopt the "3+3" principle for dose escalation until DLT is determined. The DLT observation period is 6 weeks before the induction perfusion period. This experiment will preset three dose groups: 1 × 10^12vp, 2 × 10^12vp, and 3 × 10^12vp.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): The administration cycle of this experiment includes 6 induction perfusion periods (once a week for 6 consecutive weeks) and 15 maintenance perfusion periods (once a week for the first 3 weeks after 3, 6, 12, 18, and 24 months of initial induction perfusion, for a total of 3 times a month). This study will adopt the "3+3" principle for dose escalation until DLT is determined. The DLT observation period is 6 weeks before the induction perfusion period. This experiment will preset three dose groups: 1 × 1012vp, 2 × 1012vp, and 3 × 1012vp.
  Interventions: Drug: Recombinant Human Adenovirus Type 5 injection

INTERVENTIONS:
Drug: Recombinant Human Adenovirus Type 5 injection — The administration cycle of this experiment includes 6 induction perfusion periods (once a week for 6 consecutive weeks) and 15 maintenance perfusion periods (once a week for the first 3 weeks after 3, 6, 12, 18, and 24 months of initial induction perfusion, for a total of 3 times a month). This study will adopt the "3+3" principle for dose escalation until DLT is determined. The DLT observation period is 6 weeks before the induction perfusion period. This experiment will preset three dose groups: 1 × 10^12vp, 2 × 10^12vp, and 3 × 10^12vp.

SUMMARY:
This is a prospective, open label, single center clinical study on the use of recombinant human adenovirus type 5 injection for bladder instillation therapy in high-risk non muscle invasive bladder urothelial carcinoma patients. The study was administered in a dose escalation manner, starting from a relatively safe dose of 1.0 × 10 ^ 12vp as the first dose group, and a 6-week DLT observation period was set up to ensure the safety of the study. Expected to enroll 12-18 participants. The subjects need to undergo maximum transurethral resection of the bladder (TURBT) and imaging diagnosis, and biological samples such as blood, urine, and biopsy tissue should be collected before treatment. The patient will receive bladder instillation therapy with recombinant human adenovirus type 5 injection after TURBT surgery. The subjects should receive a fixed dose of recombinant human adenovirus type 5 injection (1.0 × 10 ^ 12 vp or 2.0 × 10 ^ 12 vp or 3.0 × 10 ^ 12 vp) per week via bladder instillation for 6 weeks for induction therapy, followed by maintenance infusion of the same dose once a week for 3 weeks after the first induction infusion at 3, 6, 12, 18, and 24 months. After the first intravesical intervention for 3 months, tumor site pathology, imaging, and cytology will be obtained through diagnostic TURBT for tumor evaluation. Patients who achieve complete remission will maintain the same induction cycle, and will receive follow-up every 3 months for 2 years, every 6 months for more than 2 years, and once a year for more than 3 years. Patients who are intolerant to intravesical treatment (evaluated by the researchers) will be directly discontinued.

DETAILED DESCRIPTION:
Non muscular invasive bladder cancer (NMIBC) accounts for about 75% of all bladder malignant tumors. For NMIBC with high recurrence risk, its recurrence rate is high, about 15% -78%. The rate of progression to muscular invasion and metastasis is between 1% -45%. The long-term outcome shows that about 20% -25% of these patients will die of bladder cancer. Since the beginning of the 21st century, after obtaining positive results in many clinical trials, various oncolytic viruses have been approved for marketing both domestically and internationally.

Oncolytic viruses (including Recombinant Human Adenovirus Type 5 Injection, T-VEC, Teserpatulev, etc.) have been proven to be a promising approach for cancer treatment. The ORR of patients receiving Ankoray+chemotherapy reached 72.7%, compared to 40.3% for patients receiving chemotherapy alone. T-VEC has been used for the treatment of melanoma in Europe, the United States, and other regions. Patients receiving T-VEC have an ORR of 16.3% and a median OS of 23.3 months, while those receiving GM-CSF have an ORR of only 2.1% and a median OS of 18.9 months. Teserpaturev is based on the HSV skeleton and is used in Japan to treat glioblastoma, with a median PFS of 4.7 months and a median OS of 20.2 months, greatly changing the current treatment status.

Whether NMIBC patients can be treated with other therapies such as oncolytic virus instead of BCG has always been a hot topic in clinical research. In a phase I clinical trial consisting of 35 NMIBC patients with recurrent intravesical BCG, patients were sequentially treated with 0.1% DDM (n-dodecyl - β - D-maltoside, which can be used as a transduction enhancer) in the bladder, followed by CG0070. The CR rate was 48.6%, and the median CR time was 10.4 months. In an exploratory analysis, 81.8% of patients with critical or high Rb phosphorylation responded to treatment. The results of a subsequent phase II clinical trial (NCT02365818) showed a 6-month CR rate of 45% (95% CI 32-62%). Based on good preliminary results, the researchers initiated a phase III clinical trial (NCT04452591). The mid-term analysis data showed that the CR rate of BCG unresponsive NMIBC patients receiving CG0070 monotherapy was 75.7% (n=50/66), and the most common treatment-related adverse events in the trial included transient grade 1-2 local urogenital symptoms, with no related grade 3 or above adverse events observed. In addition, there are currently multiple NMIBC clinical trials underway for the treatment of BCG non responsiveness with oncolytic viruses.

Recombinant Human Adenovirus Type 5 Injection is an oncolytic adenovirus antitumor drug. In short, it mainly exerts anti-tumor effects through the following mechanisms: when adenovirus is infected, the E1a gene of the virus is immediately expressed to regulate the expression of other genes of the virus and promote the host cell to enter the S phase. The host cell responds by activating p53 induced apoptosis, thereby inhibiting the continued replication of the virus. At the same time, the E1b55k gene also exists in adenovirus, which can prevent E1a induced p53 effect through at least three mechanisms. Firstly, E1b55k binds to the amino terminus of p53, thereby inhibiting p53 transactivation; Secondly, E1b55k collaborates with Ad E4orf6 to hydrolyze and degrade p53 protein; Thirdly, using E1b55k alone can act as an E3 SUMO1-p53 ligase, ultimately leading to p53 polyubiquitination and proteasomal degradation. Therefore, E1b55k can counteract E1a induced p53 dependent cell apoptosis and prevent premature cell death, thereby effectively replicating the virus in normal cells. Without E1b55k, adenovirus may not be able to counteract E1a induced p53 accumulation, and therefore cannot replicate in cells with functional p53 protein. Due to the deletion or mutation of the p53 gene, p53 deficiency is common in many types of human cancers. Recombinant human adenovirus type 5 can selectively replicate in certain tumor cells by deleting fragments of E1b55k and E3 genes through gene editing, thereby achieving the effect of killing tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this clinical study, understand the study procedures, and provide written informed consent.
* Aged ≥18 years, regardless of gender.
* Eastern Cooperative Oncology Group (ECOG) performance status score ≤2.
* Expected survival time ≥2 years.
* Histologically confirmed high-risk non-muscle invasive bladder cancer (NMIBC) ("high-risk" defined in Appendix 1 ).
* No residual lesions after cystoscopy or transurethral resection of bladder tumor (TURBT) within 6 weeks prior to the first dose, or residual lesions limited to carcinoma in situ (CIS).
* Adequate Hematologic and Organ Function :

Hematologic (no blood transfusion, growth factors, or hematopoietic stimulants within 14 days):

Absolute neutrophil count (ANC) ≥1.0×10⁹/L; Platelet count (PLT) ≥100×10⁹/L; Hemoglobin (Hb) ≥80 g/L.

Liver Function :

Total bilirubin (TBIL) ≤2×ULN; Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤3×ULN.

Renal Function :

Serum creatinine (Cr) ≤1.5×ULN.

Electrocardiogram (ECG) :

QTc interval ≤450 ms (male) or ≤470 ms (female), corrected by Fridericia's formula (QTc = QT/(RR⁰·³³)).

Cardiac Ultrasound :

Left ventricular ejection fraction (LVEF) ≥50%.

Coagulation :

Activated partial thromboplastin time (APTT) ≤1.5×ULN; International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN. Contraception Requirements

* Non-sterilized participants of childbearing potential (male or female) must agree to use effective contraception (e.g., intrauterine device, oral contraceptives) during the study and for 3 months after treatment.

Female participants (or female partners of male participants) must use highly effective contraception.

* Non-sterilized female participants must have a negative serum HCG test within 7 days before the first dose and must not be lactating.

Exclusion Criteria:

* Prior Bladder Radiotherapy
* Prior Treatments Without Disease Progression (as Assessed by Investigator)
* Previous intravesical therapy with cytotoxic chemotherapy or other agents (e.g., oncolytic viruses, IL-2).
* Systemic chemotherapy, immune checkpoint inhibitors, or antibody-drug conjugates (ADCs).
* Participation in other investigational drug trials for NMIBC.
* Intravesical Bacillus Calmette-Guérin (BCG) treatment within 2 weeks before the first dose (eligible if washout period exceeds 2 weeks).
* Currently receiving investigational treatment in another clinical trial or completion of such treatment <4 weeks before the first dose in this study.
* Upper urinary tract or urethral tumors detected during screening ( CTU/MRU ). Other malignancies within 5 years before the first dose (exceptions: completely resolved carcinoma in situ or indolent malignancies like prostate cancer, per investigator's judgment).
* Active severe infections requiring IV antibiotics, antivirals, or antifungals. Grade ≥3 urinary tract infection (UTI) not recovered to Grade ≤2.
* Previous BCG therapy discontinued due to adverse events (e.g., sepsis, systemic infection, urinary incontinence) unless fully recovered to Grade ≤2 .
* Clinically Significant Cardiovascular Disease , including but not limited to:

Congestive heart failure ( NYHA Class >2 ); Unstable angina; Severe myocardial infarction within 6 months ; Symptomatic arrhythmias requiring intervention.

* Immunodeficiency or Transplant History , including HIV-positive serology and other acquired/congenital immunodeficiencies.
* History of organ transplantation or current immunosuppressant use.
* Active Viral Hepatitis Hepatitis B : HBeAg-positive and HBV DNA ≥500 IU/mL. Hepatitis C : Anti-HCV-positive and HCV RNA above the lower limit of detection.

Hypersensitivity or Intolerance

* Known allergy or intolerance to the study drug or its excipients.
* Any other severe physical/psychiatric illness, abnormal lab results, or factors that may: Increase study participation risks; Interfere with study results; Investigator's discretion for ineligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
3-month CR | 3 months
  Complete response (CR) rate of patients receiving bladder instillation of recombinant human adenovirus type 5 injection at 3 months in each dose group.CR is defined as negative urine cytology examination, no tumor detected on imaging, and negative biopsy in the ITT population. Subjects with no response data in the primary analysis population (FAS) will be counted as non responders. Analyze based on the effectiveness analysis set
DLT | 6 weeks
  DLT is defined as any of the following events related to the study drug that occur during the DLT observation period (grading criteria refer to NCI CTCAE 5.0):
  1. Hematological toxicity:
     * Grade 4 neutrophil count decrease lasting>5 days;
       -≥ Grade 3 febrile neutropenia;
     * Grade 4 anemia;
     * Grade 4 platelet count decreased;
     * Grade 3 platelet count decrease lasting>7 days;
     * Grade 3 platelet count decrease accompanied by significant clinical bleeding symptoms;
     * The decrease in lymphocyte count at level 4 lasts for ≥ 14 days.
  2. Liver toxicity:
     * Level 4 ALT or AST elevation;
     * Level 3 ALT or AST elevation accompanied by ≥ level 2 TBIL elevation;
  3. Urinary tract related adverse reactions:
     -Bladder perforation or urinary fistula;
     -≥ grade 3 urinary tract infection, bladder spasm, cystitis, hematuria, urinary retention, urinary pain, urinary incontinnence, and lasted for>7 days after symptomatic treatment.
  4. Other non hematological toxicities:
     * Other non hematological toxicities of grade ≥ 3.
MTD | 6 weeks
  This study will adopt dose escalation, starting from the initial dose group, with at least 3 cases in each dose group. If no DLT occurs, it will be raised to the next dose group; If one case of DLT occurs, three cases will be re enrolled in the same dose group. If the three newly enrolled cases do not have DLT, they will be promoted to the next dose group. Otherwise, the dose escalation experiment will be stopped. This dose level is the MTD

SECONDARY OUTCOMES:
AEs | 12 months
  The types, incidence, severity (rated according to CTCAE v5.0), duration, and correlation with the investigational drug of adverse events (AEs) and serious adverse events (SAEs), including vital signs, abnormal electrocardiograms, and laboratory tests;
DoR | 24 months
  Duration of CR remission
6-month CR | 6 months
12-month CR | 12 months
RFS | 24 months
  relapse-free survival
BI-EFS | 24 months
  Event free survival with intact bladder
Time to Cystectomy | 24 months
  The time from the end of medication to bladder resection
Radical cystectomy rate | 24 months

OTHER OUTCOMES:
Biomarkers | 12 months
  Biomarkers of tissue, blood, and urine, including but not limited to CCF, CNA, and other parameters of utDNA, before and during the infusion of recombinant human adenovirus type 5 injection
Drug Recovery in Instillation Fluid and Urine | 12 months
PK parameter | 12 months
  Pharmacokinetic parameters including plasma drug concentration , etc.
PD parameter | 12 months
  Including but not limited to levels of cytokines such as interleukin-6 (IL-6) and interferon-I (IFN-I) in urine
Immunogenicity | 12 months
  Including the occurrence of positive results for drug-resistant antibodies and neutralizing antibodies.